CLINICAL TRIAL: NCT03838757
Title: Maximal Exercise Capacity, Extra-pulmonary Characteristics and Physical Activity Levels in Patients With Lung Cancer With Complete Remission .
Brief Title: Maximal Exercise Capacity and Extra-pulmonary Characteristics in Patients With Lung Cancer With Complete Remission .
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate Professor, Gazi University
Other Study IDs: Gaziuniversity13
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Exercise capacity; Cardiopulmonary exercise test; Respiratory muscle strength; Physical activity; Pulmonary functions; Peripheral Muscle Strength; Quality of life; Sleep of quality; Dyspnea; Depression; Fatigue; Cough
MeSH Terms: conditions — Lung Neoplasms; Motor Activity; Dyspnea; Depression; Fatigue; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Maximal exercise capacity was assessed using cardiopulmonary exercise testing (CPET), exercise capacity six minute walk test, physical activity multi-sensor activity monitor, pulmonary function spirometry, respiratory muscle strength mouth pressure device, peripheral muscle strength hand held dynamometer, dyspnea Modified Medical Research Council Dyspnea Scale (MMRC), fatigue Fatigue Severity Scale, quality of life The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) and Functional Assessment of Cancer Therapy - Lung cancer quality of life questionnaire (FACT-L), depression Montgomery Asberg Depression scale, sleep of quality Pittsburgh Sleep Quality index and cough using Leicester Cough Questionnaire were evaluated.
- Healthy controls: Maximal exercise capacity was assessed using cardiopulmonary exercise testing (CPET), exercise capacity six minute walk test, physical activity multi-sensor activity monitor, pulmonary function spirometry, respiratory muscle strength mouth pressure device, peripheral muscle strength hand held dynamometer, dyspnea Modified Medical Research Council Dyspnea Scale (MMRC), fatigue Fatigue Severity Scale, quality of life The European Organization for Research and Treatment of Cancer quality of life questionnaire (EORTC QLQ-C30) and Functional Assessment of Cancer Therapy - Lung cancer quality of life questionnaire (FACT-L), depression Montgomery Asberg Depression scale, sleep of quality Pittsburgh Sleep Quality index and cough using Leicester Cough Questionnaire were evaluated.

SUMMARY:
While lung cancer are rare disease in the early 20th century, its incidence increased in parallel with the increase in smoking habits. It is the most common type of cancer in the world. Despite advances in the efficacy of chemotherapy and radiotherapy regimens, surgical resection is the most effective curative treatment modality to improve survival in non-small cell lung cancer. Pulmonary resection candidates are selected according to not only tumor type and stage, but also functional status, exercise capacity, underlying lung disorders and health-related quality of life assessments. Patients with lung cancer often have lung and heart comorbidities that affect the outcome of the outcome measures and restricts cancer treatment options. In patients with lung cancer, shortness of breath, physical inactivity, weakness in peripheral muscles and exercise intolerance are described. Pulmonary rehabilitation is a multidisciplinary treatment designed to improve exercise capacity, functional status, health-related quality of life and to reduce the attenuation of chronic shortness of breath and fatigue in patients with chronic lung problems.

In literature, the effect of surgery in patients with lung cancer on postoperative respiratory muscle strength is not clear. There is no study investigating the effect of chemotherapy and radiotherapy on respiratory muscle strength. For these reasons, the aim of the study was to evaluate the curative period of non-small cell lung cancer patients with reliability and validity assessment methods. The hypothesis of our study was; when compared with patients with lung cancer and healthy individuals, exercise capacity, respiratory and peripheral muscle strength, physical activity levels, sleep and quality of life of lung cancer patients are reduced; dyspnoea, fatigue, depression, cough and pain levels increase.

DETAILED DESCRIPTION:
According to sample size calculation 20 lung with complete remission cancer patients and 20 healthy individuals were included in the study. Cross-sectional observational research. The demographic, physical and physiological characteristics were recorded from the patient files. Exercise capacity (using cardiopulmonary exercise testing), physical activity, pulmonary functions, respiratory and peripheral muscle strength, dyspnea and fatigue perception, depression, cough, pain and quality of life were evaluated. Primary outcome measurement is maximal exercise capacity. Secondary outcomes are respiratory and peripheral muscle strength, pulmonary functions, physical activity, dyspnea and fatigue perception, depression, cough, pain and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with; Diagnosed with lung cancer Stage 1, stage 2 and stage 3 patients in lung cancer patients Clinically stable and Under standard medication patients were included.

Exclusion Criteria:

* Patients with Metastasis Orthopedic and neurological problems Acute infection Non-co-operable
* Healthy Subjects with Any diagnosed disease were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with lung cancer were included in the patients group and 20 healthy individuals were included in the control group
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | Second day
  Cardiopulmonary exercise testing (Oxygen consumption measurement during test).

SECONDARY OUTCOMES:
Functional exercise capacity | First day
  The six-minute walking test (6-MWT) was used to evaluate submaximal exercise capacity.
Physical activity | First day
  Physical activity will be evaluated multi sensor activity monitor for 2 consecutive days.
Pulmonary function test | First day
  This test was evaluated using a spirometry by which is evaluated dynamic lung functions expressed as percentages of expected values.
Inspiratory and Expiratory muscle strength (MIP, MEP) | First day
  Respiratory muscle strength was evaluated with a mouth pressure device
Peripheral muscle strength | First day
  Peripheral muscle strength was evaluated with a hand-held dynamometer.
Dyspnea | First day
  The severity of dyspnea during daily living activities was evaluated using the Modified Medical Research Council (MMRC) dyspnea scale. Dyspnea is graded as follows: zero (dyspnea only with strenuous exercise), one (dyspnea when hurrying or walking up a slight hill), two (walks slower than people of the same age due to dyspnea or having to stop for breath when walking at own pace), three (stops for breath after walking 100 yards or after a few minutes) and four (too dyspneic to leave house or breathless when dressing). The minimal clinically important difference (MCID) is 1 unit for the MMRC dyspnea scale.
Fatigue Severity | First day
  The Turkish version of Fatigue Severity Scale, which is a valid and reliable test, was performed to the recipients for evaluation of fatigue severity. Self-administered questionnaire is comprised of nine questions. The average score is identified on seven-point scale. Patients select a number from 1 to 7 for each 9 questions which demonstrates from strong disagreement to strong agreement, respectively. The cut-off score for fatigue severity is 36 according to this scale, if the total score obtained from this scale is higher than 36, the recipient is defined as severe fatigue.
Life Quality | First day
  Quality of life was measured using Turkish version of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 version 3.0 (EORTCQLQ) which is widely used as health related quality of life questionnaire in cancer patients. The cancer-specific questionnaire has 30 questions and incorporates five functional scales, three symptom scales, a global health status and several single items. All item scores are transformed to 0-100. Higher values indicate higher functional/healthy level in functional scales, a higher quality of life level in global health status and increased symptoms in symptom scales.
Depression | First day
  Montgomery Asberg Depression Rating Scale (MADRS) (Turkish version of scale) This assessment tool contains 10 items with a score from 0 to 6, thus the maximum score is 60. A higher score indicates a more severe depression.
Sleep of quality | First day
  Sleep quality of the individuals was evaluated with the Turkish version of Pittsburgh Sleep Quality Index. It is an individual evaluation scale that evaluates sleep quality and sleep disturbance in the last one month period.
Cough | First day
  The Turkish version of the Leicester Cough Scale (LÖQ) was used to assess the health-related quality of life of individuals with chronic cough. The scale evaluates chronic cough consisting of 19 items, including physical (8 items), psychosocial (7 items) and social (4 items) subsections. Each item is scored between 1 (always) and 7 (never). The total score is 3-21 points. The high scores obtained from this questionnaire, which evaluates the effect of the symptoms that have been going on for the last two weeks, show less impact on cough and lower scores indicate more impact.
Life Quality | Second day
  Functional Assessment of Cancer Therapy - Lung cancer Quality of life questionnaire (Turkish version) is used to assess the quality of life of lung cancer patients from many cultures all over the world. It is an individual applied scale and consists of 36 questions specific to lung cancer. Body is a scale consisting of 5 subsections including status, social life and family situation, emotional state, activity status and other concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Pelin Dündar, MSc, Study Chair — Gazi University; Meral Boşnak Güçlü, Assoc. Prof, Study Director — Gazi University; Aydın Çiltaş, MD, Principal Investigator — Gebze Medical Park Hospital; Mustafa Benekli, MD, Principal Investigator — Cukurambar/Ankara
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Yenimahalle, Turkey (Türkiye)

REFERENCES:
- [Result] Cavalheri V, Jenkins S, Cecins N, Gain K, Phillips M, Sanders LH, Hill K. Impairments after curative intent treatment for non-small cell lung cancer: a comparison with age and gender-matched healthy controls. Respir Med. 2015 Oct;109(10):1332-9. doi: 10.1016/j.rmed.2015.08.015. Epub 2015 Aug 29. PMID 26342839
- [Result] Granger CL, Denehy L, Parry SM, Martin J, Dimitriadis T, Sorohan M, Irving L. Which field walking test should be used to assess functional exercise capacity in lung cancer? An observational study. BMC Pulm Med. 2015 Aug 12;15:89. doi: 10.1186/s12890-015-0075-2. PMID 26264470
- [Result] Cavalheri V, Jenkins S, Cecins N, Gain K, Hill K. Comparison of the six-minute walk test with a cycle-based cardiopulmonary exercise test in people following curative intent treatment for non-small cell lung cancer. Chron Respir Dis. 2016 May;13(2):118-27. doi: 10.1177/1479972316631137. Epub 2016 Feb 11. PMID 26869579
- [Result] Granger CL, Parry SM, Edbrooke L, Denehy L. Deterioration in physical activity and function differs according to treatment type in non-small cell lung cancer - future directions for physiotherapy management. Physiotherapy. 2016 Sep;102(3):256-63. doi: 10.1016/j.physio.2015.10.007. Epub 2015 Oct 23. PMID 26597694
- [Result] Arbane G, Douiri A, Hart N, Hopkinson NS, Singh S, Speed C, Valladares B, Garrod R. Effect of postoperative physical training on activity after curative surgery for non-small cell lung cancer: a multicentre randomised controlled trial. Physiotherapy. 2014 Jun;100(2):100-7. doi: 10.1016/j.physio.2013.12.002. Epub 2014 Feb 12. PMID 24703523
- [Result] Hashmi A, Baciewicz FA Jr, Soubani AO, Gadgeel SM. Preoperative pulmonary rehabilitation for marginal-function lung cancer patients. Asian Cardiovasc Thorac Ann. 2017 Jan;25(1):47-51. doi: 10.1177/0218492316683757. Epub 2016 Dec 5. PMID 27913735